CLINICAL TRIAL: NCT00640185
Title: A Pilot, Randomized, Double-Blind, Placebo-Controlled, Parallel-Group, Phase 2 Study of the Safety, Tolerability and Efficacy of 40 mg QD and 80 mg QD ABT-089 in Adults With Attention Deficit-Hyperactivity Disorder (ADHD)
Brief Title: Safety, Tolerability and Efficacy Study of ABT-089 in Adults With Attention-Deficit/Hyperactivity Disorder (ADHD)
Status: Completed | Phase: Phase 2 | Type: Interventional
Sponsor: AbbVie (prior sponsor, Abbott) (Industry)
Responsible Party: Sponsor
Organization: AbbVie (Industry)
Allocation: Randomized | Model: Parallel | Masking: Triple | Purpose: Treatment
Other Study IDs: M10-346
Record Dates: First submitted 2008-03-18; First posted 2008-03-21 (Estimated); Last update posted 2013-01-18 (Estimated); Status verified 2013-01

CONDITIONS: Attention-Deficit/Hyperactivity Disorder
MeSH Terms: conditions — Attention Deficit Disorder with Hyperactivity | interventions — pozanicline

STUDY DESIGN:
Who Masked: Participant, Care Provider, Investigator
Oversight: Data Monitoring Committee: No

ARMS (3):
- 1 (Placebo Comparator)
  Interventions: Drug: ABT-089; Drug: Placebo
- 2 (Experimental)
  Interventions: Drug: ABT-089; Drug: Placebo
- 3 (Experimental)
  Interventions: Drug: ABT-089; Drug: Placebo

INTERVENTIONS:
Drug: ABT-089 — Subjects will take up to two 40 mg tablets once daily for 8 weeks.
Drug: Placebo — Subjects will take one or two placebos once daily for the duration of the study.

SUMMARY:
The purpose of this study is to test if the investigational medication ABT-089 is a safe and effective treatment for adults with Attention-Deficit/Hyperactivity Disorder (ADHD).

ELIGIBILITY:
Inclusion Criteria:

* Have voluntarily signed an informed consent form.
* Meet diagnostic criteria for attention-deficit/hyperactivity disorder (ADHD) based on detailed evaluation and interview with subject.
* Subject is generally in good health based on medical history, physical examination, clinical lab tests and ECG.
* Female subjects of child-bearing potential must have a negative urine pregnancy test at screening and baseline and agree to comply with applicable contraceptive requirements.
* Male subjects must agree to comply with applicable contraceptive requirements.
* Subject is able to keep required appointments for clinic visits and all tests, including blood draws and examinations.

Exclusion Criteria:

* Subject has a current or past diagnosis of schizoaffective disorder, schizophrenia, obsessive-compulsive disorder, drug-induced psychosis, bipolar disorder, psychotic disorder.
* Current diagnosis of major depressive disorder, generalized anxiety disorder, PTSD or has a sleep disorder requiring treatment of any kind.
* Subject has a history of, or ongoing, serious medical problem.
* Subject has a history of significant allergic reaction to any drug.
* Subject is planning to begin any type of behavioral or psychotherapy for treatment of ADHD.
* Subject requires ongoing treatment with any psychiatric medication.

Ages: 18 Years to 60 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult
Enrollment: 160 (Actual)
Dates: Start 2008-03; Primary Completion 2008-08 (Actual); Study Completion 2008-08 (Actual)

PRIMARY OUTCOMES:
CAARS: Inv Total Score | Screening, Day -1, Day 7, Day 14, Day 28, Day 42 and Day 56

SECONDARY OUTCOMES:
CAARS Inattentive and Hyperactive/Impulsivity Sub-scale scores, CAARS ADHD Index, CGI-ADHD-S, AISRS, CAARS:Self | Screening, Day -1, Day 7, Day 14, Day 28, Day 42 and Day 56
TASS, AAQoL, WPAI | Day -1, Day 28, Day 56
BRIEF-A, FTND | Day-1, Day 56
QSU-Brief, Number of Cigarettes smoked per day | Day -1, Day 7, Day 14, Day 28, Day 42, Day 56

CONTACTS AND LOCATIONS:
Overall Officials: Earle Bain, Study Director — AbbVie
Locations (12):
- United States (12):
  - Site Reference ID/Investigator# 7546, Lafayette, California
  - Site Reference ID/Investigator# 7551, Jacksonville, Florida
  - Site Reference ID/Investigator# 7553, Orlando, Florida
  - Site Reference ID/Investigator# 7545, Overland Park, Kansas
  - Site Reference ID/Investigator# 7552, Farmington Hills, Michigan
  - Site Reference ID/Investigator# 7548, Troy, Michigan
  - Site Reference ID/Investigator# 7554, Eugene, Oregon
  - Site Reference ID/Investigator# 7547, Portland, Oregon
  - Site Reference ID/Investigator# 7555, Memphis, Tennessee
  - Site Reference ID/Investigator# 7549, Virginia Beach, Virginia
  - Site Reference ID/Investigator# 7550, Bellevue, Washington
  - Site Reference ID/Investigator# 7631, Seattle, Washington

REFERENCES:
- [Derived] Bain EE, Apostol G, Sangal RB, Robieson WZ, McNeill DL, Abi-Saab WM, Saltarelli MD. A randomized pilot study of the efficacy and safety of ABT-089, a novel alpha4beta2 neuronal nicotinic receptor agonist, in adults with attention-deficit/hyperactivity disorder. J Clin Psychiatry. 2012 Jun;73(6):783-9. doi: 10.4088/JCP.10m06719. PMID 22795204